CLINICAL TRIAL: NCT00793416
Title: Accuracy of ShuntCheck and MRI in Detection of Shunt Obstruction in Patients Receiving Shunt Patency Test
Brief Title: ShuntCheck Accuracy in Detecting Shunt Obstruction Normal Pressure Hydrocephalus (NPH) Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Loss of study staffing
Sponsor: NeuroDx Development (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NDX01-22-2003
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Normal Pressure Hydrocephalus; Valve Adjustment; Blocked Shunt in NPH patients; Diagnosis of blockage
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ShuntCheck measure (Experimental): All patients will have ShuntCheck measurements along with radionuclide shunt patency testing.
  Interventions: Device: Shunt flow detection

INTERVENTIONS:
Device: Shunt flow detection — Shunt flow detection based upon ShuntCheck results compared to radionuclide test results

SUMMARY:
The purpose of this study is to examine the role of ShuntCheck and MR Imaging in evaluating the presence or absence of Shunt Obstruction in the patients of Hydrocephalus or Idiopathic Intracranial Hypertension (IIH) undergoing radionuclide test for suspected shunt obstruction. This is an exploratory study to determine how a non-invasive device can assist in detection of presence of flow in these patients.

DETAILED DESCRIPTION:
This study aims to correlate findings of ShuntCheck and MRI with the Radionuclide patency study. Patients will be enrolled if they have Hydrocephalus or IIH, present with symptoms of shunt obstruction and will need to undergo shunt patency test and an MRI along with standard of care radionuclide study. The ShuntCheck study will be conducted in a clinic, doctor's office or in an emergency room by the treating physician or by trained health care professionals.

Also, patients who are found with shunt obstruction as diagnosed by Radionuclide study will undergo shunt revision and the findings of the study will be correlated with operative findings. Post Shunt replacement patients who also receive adjustable valve will be evaluated with shunt Check, before and after adjustment of valves to detect changes in flow as detected by shunt check.

This is an exploratory study to determine how a non-invasive device can assist in detection of presence of flow in these patients.

Approximately 20 subjects will be enrolled in a single site in this proof of concept, physician sponsored study. An approved, commercial device will be available to the site prior to start of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients > 35 years capable and willing to consent for their participation or consent obtained from a legal guardian.
2. Patients with an indwelling shunt and clinical assessment strongly suggestive of shunt obstruction
3. Patients are candidates for shunt patency procedures in the elective extension

Exclusion Criteria:

1. Patients <35 years of age
2. Patients with symptoms attributable to valve malfunction or shunt infection
3. Patients who need urgent shunt replacement and therefore cannot wait for the SHUNTCHECK evaluation of shunt patency.
4. Patients with edema or wound of skin overlying the shunt tissue.
5. Patients not capable or not willing to consent to participate in the study

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Exploratory Evaluation of the Utility of ShuntCheck in detection of ShuntFlow in patients admitted with potential shunt obstruction | Pre and post shunt revision surgery

SECONDARY OUTCOMES:
To assess any adverse events that arise from conducting ShuntCheck test To assess the cost effectiveness of ShuntCheck screening upon completion of the study | Pre and post shunt revision surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Rigamonti, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Medical Center, Baltimore, Maryland, United States